CLINICAL TRIAL: NCT07368426
Title: Immediate Effects of Strain Counterstrain Versus Fascial Distortion Model on Pain and Function in Individuals With Latent Myofascial Trigger Points of the Upper Trapezius: A Pilot Study
Brief Title: Immediate Effects of Strain Counterstrain Versus Fascial Distortion Model on Upper Trapezius Latent Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungnam University (Other)
Responsible Party: Principal Investigator, JiYoung Kim, Adjunct Professor, Physical Therapy, Kyungnam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JYK-2025-02
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Latent Myofascial Trigger Points; Upper Trapezius Muscle
Keywords: Strain Counterstrain; Fascial Distortion Model; Manual Therapy; Myofascial Trigger Point; Upper Trapezius

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strain Counterstrain Group (Experimental): Participants received a single session of strain counterstrain manual therapy applied to latent myofascial trigger points of the upper trapezius muscle.
  Interventions: Other: Strain Counterstrain
- Fascial Distortion Model Group (Experimental): Participants received a single session of fascial distortion model manual therapy applied to latent myofascial trigger points of the upper trapezius muscle.
  Interventions: Other: Fascial Distortion Model

INTERVENTIONS:
Other: Strain Counterstrain — Strain counterstrain is an indirect manual therapy technique in which the body is passively positioned in a pain-free posture to reduce nociceptive input and muscle tension. In this study, a single session of strain counterstrain was applied to latent myofascial trigger points of the upper trapezius muscle.
  Arms: Strain Counterstrain Group
Other: Fascial Distortion Model — The fascial distortion model is a direct manual therapy approach that applies localized, high-intensity pressure to specific fascial distortions identified through patient body language and palpation. In this study, a single session of fascial distortion model intervention was applied to latent myofascial trigger points of the upper trapezius muscle.
  Arms: Fascial Distortion Model Group

SUMMARY:
This pilot study aimed to compare the immediate effects of two manual therapy techniques, strain counterstrain (SCS) and the fascial distortion model (FDM), on pain-related outcomes and neuromuscular function in individuals with latent myofascial trigger points of the upper trapezius muscle. Twenty healthy adults with identified latent trigger points were randomly assigned to receive a single session of either SCS or FDM. Cervical range of motion, proprioception, pressure pain threshold, and cervical muscle strength were assessed before and immediately after the intervention. This study was conducted to obtain preliminary data regarding the short-term effects of two manual therapy approaches with contrasting stimulation characteristics.

DETAILED DESCRIPTION:
Musculoskeletal pain of the cervical region is a prevalent health problem, and the upper trapezius muscle is frequently involved due to postural overload and mechanical stress. These factors are commonly associated with the development of latent myofascial trigger points, which may restrict range of motion and impair neuromuscular function even in the absence of spontaneous pain.

Various manual therapy techniques have been used to manage myofascial trigger points. Strain counterstrain (SCS) is an indirect, low-intensity technique that aims to reduce nociceptive input and muscle spindle activity by positioning the body in a pain-free posture. In contrast, the fascial distortion model (FDM) is a direct manual therapy approach that applies relatively high-intensity pressure to specific fascial distortions identified through patient body language and palpation.

This study was designed as a pilot, parallel-group, pre-post comparative trial to explore the immediate effects of SCS and FDM on pain-related and neuromuscular outcomes in individuals with latent myofascial trigger points of the upper trapezius. Twenty healthy adults were randomly assigned to receive a single session of either SCS or FDM. Cervical range of motion, joint position error, pressure pain threshold, and cervical muscle strength were assessed before and immediately after the intervention. The findings of this study are intended to provide preliminary evidence to inform future large-scale clinical trials comparing manual therapy techniques with differing stimulation characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 39 years.
* Presence of latent myofascial trigger points in the upper trapezius muscle.
* No history of neurological or orthopedic disorders within the past six months.
* Willingness to participate and provision of written informed consent.

Exclusion Criteria:

* Current or previous complaints of neck or shoulder pain.
* Ongoing treatment for musculoskeletal conditions.
* History of physical therapy or chiropractic treatment within the past six months.
* History of surgery or trauma involving the head or upper trunk.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Cervical Range of Motion | Before and immediately after the intervention
  Active cervical range of motion was measured using a Cervical Range of Motion (CROM) device in flexion, extension, lateral flexion, and rotation.
Pressure Pain Threshold | Before and immediately after the intervention
  Pressure pain threshold at the latent myofascial trigger point of the upper trapezius muscle was measured using a digital algometer.

SECONDARY OUTCOMES:
Cervical Proprioception | Before and immediately after the intervention
  Cervical proprioception was assessed using joint position error during cervical lateral flexion measured with a CROM device.
Cervical Muscle Strength | Before and immediately after the intervention
  Isometric cervical muscle strength was measured using a digital muscle tester during flexion, extension, lateral flexion, and rotation.

CONTACTS AND LOCATIONS:
Overall Officials: JiYoung Kim, PT, PhD, Principal Investigator — Kyungnam University
Locations (1):
- Kyungnam University, Changwon, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No